CLINICAL TRIAL: NCT06563388
Title: (ID-COMET) A Randomized Phase III Trial of Immediate Versus Six-Month Delayed Comprehensive Treatment of 1-10 Oligometastatic Tumors With or Without Synchronous Primary
Brief Title: Stereotactic Ablative Radiotherapy (SABR) for the Treatment of Patients With Metastatic Cancer, ID-COMET Trial
Acronym: ID-COMET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-3739023
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Oligometastasis; Lung Cancer; Colo-rectal Cancer; Prostate Cancer
MeSH Terms: conditions — Lung Neoplasms; Colonic Neoplasms; Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard Therapy followed by SABR - Trial 1-3 Arm 1 (Experimental)
  Interventions: Procedure: Stereotactic Ablative Radiotherapy; Other: Best Practice
- SABR plus Standard therapy - Trial 1-3 Arm 2 (Experimental)
  Interventions: Procedure: Stereotactic Ablative Radiotherapy; Other: Best Practice
- Trial 4 - Immediate SABR plus standard of care (Experimental)
  Interventions: Procedure: Stereotactic Ablative Radiotherapy; Other: Best Practice

INTERVENTIONS:
Procedure: Stereotactic Ablative Radiotherapy — Radiation therapy begins after 3 months of Standard of care
  Other Names: SABER; SABR/SBRT
Other: Best Practice — Receive standard of care therapy
  Other Names: Standard of Care

SUMMARY:
This protocol is comprised of three unblinded, randomized, single-center studies to evaluate the impact of immediate versus three-month delayed comprehensive ablative treatment on survival in newly diagnosed metastatic patients with lung (Trial 1), colorectal (Trial 2), and prostate (Trial 3) cancers

ELIGIBILITY:
Inclusion Criteria:

* Age 1 year or older.
* Willing to provide informed consent.
* ECOG ≤ 3.
* Life expectancy > 6 months.
* Trials 1-3: Histologically confirmed lung, prostate or colorectal malignancy with metastatic disease detected on imaging. Biopsy of metastasis is preferred, but not required.
* Trial 4: Any malignancy with metastasis. Participants with liquid tumors are eligible provided they have biopsy confirmed refractory disease and are eligible for salvage radiotherapy.
* Newly diagnosed metastatic (1-10 sites)patients for Trials 1-3. Previously diagnosed metastatic patients (1-10 sites or oligoprogression in 5 or fewer sites with no limit on total number for Trial 4.
* Restaging completed within 12 (+/- 4) weeks prior to randomization.

  * For patients receiving thoracic radiotherapy, the enrolling physician must confirm there are no computed tomography (CT) changes suggestive of fibrotic interstitial lung disease (ILD) (i.e., reticular changes, traction bronchiectasis, or honeycombing) reported on any prior CT scans. If any are present, the patient must be assessed by a respirologist to rule out ILD prior to enrollment.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry.

Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* . Participants who have no option for standard systemic therapy or refuse systemic therapy.
* Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
* Serious medical comorbidities precluding radiotherapy. These include ILD in patients requiring thoracic radiation, Crohn's disease in patients where the gastrointestinal (GI tract will receive radiotherapy, or ulcerative colitis where the bowel will receive radiotherapy and connective tissue disorders such as lupus or scleroderma.
* For patients with liver metastases, moderate/severe liver dysfunction (Child Pugh B or C); please see the Child-Pugh score calculator.
* Substantial overlap with a previously treated radiation volume. Prior radiotherapy in general is allowed, as long as the composite plan meets dose constraints herein. For patients treated with radiation previously, biological effective dose calculations should be used to equate previous doses to the tolerance doses listed in Appendix E. All such cases must be discussed with the PI or Co-I .

  * Malignant pleural effusion.
* Inability to treat all sites of disease.

  * Metastatic disease that invades any of the following: GI tract (including esophagus, stomach, small or large bowel) or skin.
  * Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
  * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
  * Pregnant or nursing female participants.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2032-09-18 (Estimated); Study Completion 2032-09-18 (Estimated)

PRIMARY OUTCOMES:
Overall Survival - Trial 1 and 2 | UP to 5 years
  Calculated from the time of randomization until death
Androgen DeprivationTherapy (ADT)-free survival - Trial 3 | Up to 5 years
  The time from radomization until receipt of ADT, death due to any cause, end of study or last follow up.

SECONDARY OUTCOMES:
Change in Quality of Life | Up to 5 years after radiation treatment
  Quality of life will be assessed using The EORTC Core Quality of Life questionnaire (EORTC-QLC30). This questionnaire measures cancer patients' physical, psychological and social functions. This 30 item questionnaire ranges from 1 (not at all ) to 4 (Very much) except for the global health status/quality-of-life scale, which has response options ranging from (1) "very poor" to (7) "excellent"
Physician determined Radiation related toxicity | 5 years
  To document toxicity in patients using the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 5 for each organ treated

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States